CLINICAL TRIAL: NCT05164094
Title: A Phase 1/2, Randomized, Observer-Blind, Placebo-Controlled, Dose-Ranging Study of an Epstein-Barr Virus (EBV) Candidate Vaccine, mRNA-1189, in 10- to 30-Year-Old Healthy Adolescents and Adults
Brief Title: A Study of an Epstein-Barr Virus (EBV) Candidate Vaccine, mRNA-1189, in 10- to 30-Year-Old Healthy Adolescents and Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1189-P101
Record Dates: First submitted 2021-12-01; First posted 2021-12-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Epstein-Barr Virus Infection
Keywords: Infectious mononucleosis; Mononucleosis
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infectious Mononucleosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A: mRNA-1189 Dose Level 2 (Experimental): Participants will receive 3 intramuscular (IM) injections of mRNA-1189 at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part A: mRNA-1189 Dose Level 3 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part A: mRNA-1189 Dose Level 4 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 4 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part A: Placebo (Placebo Comparator): Participants will receive 3 IM injection of study drug-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo
- Part B: mRNA-1189 Dose Level 1 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part B: mRNA-1189 Dose Level 2 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part B: mRNA-1189 Dose Level 3 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part B: mRNA-1189 Dose Level 4 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 4 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part B: Placebo (Placebo Comparator): Participants will receive 3 IM injection of study drug-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo
- Part C: mRNA-1189 Dose Level 1 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 1 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part C: mRNA-1189 Dose Level 2 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 2 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part C: mRNA-1189 Dose Level 3 (Experimental): Participants will receive 3 IM injections of mRNA-1189 at Dose Level 3 on Days 1, 57, and 169.
  Interventions: Biological: mRNA-1189
- Part C: Placebo (Placebo Comparator): Participants will receive 3 IM injection of study drug-matching placebo on Days 1, 57, and 169.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1189 — Sterile liquid for injection
  Arms: Part A: mRNA-1189 Dose Level 2; Part A: mRNA-1189 Dose Level 3; Part A: mRNA-1189 Dose Level 4; Part B: mRNA-1189 Dose Level 1; Part B: mRNA-1189 Dose Level 2; Part B: mRNA-1189 Dose Level 3; Part B: mRNA-1189 Dose Level 4; Part C: mRNA-1189 Dose Level 1; Part C: mRNA-1189 Dose Level 2; Part C: mRNA-1189 Dose Level 3
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo

SUMMARY:
The main objective of Part A of this trial is to evaluate the safety and reactogenicity of mRNA-1189 in 18- to 30-year-old healthy adults, the main objective of Part B is to evaluate the safety and reactogenicity of mRNA-1189 in 12- to <18-year-old healthy EBV-seronegative adolescents, and the main objective of Part C is to evaluate the safety and reactogenicity of mRNA-1189 in 10- to 21-year-old healthy adolescents and adults.

ELIGIBILITY:
Inclusion Criteria:

* According to the assessment of the investigator, is in good general health and can comply with study procedures.

Part A: Healthy adult from 18 to 30 years of age (inclusive) at the time of consent (Screening Visit, Day 0).

Part B:

Healthy baseline EBV-seronegative adolescents from 12 to <18 years of age at the time of consent (Screening Visit, Day 0).

Part C:

Healthy adolescents and adults from 10 to 21 years of age (inclusive) at the time of consent (Screening Visit, Day 0).

Exclusion Criteria:

* Has had significant exposure to someone with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or COVID-19 in the past 14 days prior to the screening visit, if the participant has not been fully vaccinated against COVID-19 at least 14 days prior to the screening visit.
* Has symptomatic acute or chronic illness requiring ongoing medical or surgical care, to include changes in medication in the past 2 months indicating that chronic illness/disease is not stable (at the discretion of the investigator).
* Significant, progressive, unstable or uncontrolled clinical condition, including any condition that may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures per investigator judgement.
* Has a history of myocarditis, and/or pericarditis.
* Has received or plans to receive any licensed or authorized vaccine, to include COVID-19 vaccines, ≤28 days prior to the first injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after any study vaccine injection, with the exception of licensed influenza vaccines, which may be received more than 14 days before or after any study vaccine injection.

Note: Other inclusion and exclusion criteria may apply.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 867 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 176 (7-day follow-up after vaccination)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 197 (28-day follow-up after vaccination)
Number of Participants with SAEs, MAAEs, Any AEs Leading to Withdrawal From Study/Discontinuation of Study Vaccine and AEs of Special Interest (AESIs) | Day 1 to end of study (EOS) (Day 505)
Number of Participants with Laboratory Abnormalities | Up to Day 176 (7-day follow-up after vaccination)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of B-Cell Neutralizing Antibody (nAb) and/or Antigen-Specific Binding Antibody (bAb) | Days 1, 85, and 197
Geometric Mean Fold Rise (GMFR) of B-Cell nAb and Antigen-Specific bAb | Days 1, 85, and 197
Number of Participants With Seroconversion of B-Cell nAbs and/or Antigen-Specific bAbs | Days 1, 85, and 197
  The number of initially EBV-negative participants with seroconversion from below the lower limit of quantification (LLOQ) to above the LLOQ for EBV-specific (vaccine antigen) binding and nAbs responses and the initially EBV-positive participants with > 2-, 3-, and 4-fold increases in serum binding or nAb titers from baseline (if above LLOQ) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (64):
  - Medical Affiliated Research Institute, Huntsville, Alabama
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Smart Cures Clinical Research, Anaheim, California
  - Benchmark Research - Colton - HyperCore - PPDS, Colton, California
  - Fomat Medical Research, Oxnard, California
  - Center For Clinical Trials LLC -Paramount, Paramount, California
  - Artemis Institute For Clinical Research LLC - Riverside - Headlands - PPDS, Riverside, California
  - Peninsula Research Associates - Headlands Research - PPDS, Rolling Hills, California
  - Velocity Clinical Research - Banning - PPDS, San Bernardino, California
  - Acclaim Clinical Research, San Diego, California
  - California Research Foundation - 4180 Ruffin Rd, San Diego, California
  - Orange County Research Center, Tustin, California
  - Research Centers of America - ERG, Hollywood, Florida
  - Jacksonville Center For Clinical Research - ERN - PPDS, Jacksonville, Florida
  - iResearch Savannah - CenExel - PPDS, Savannah, Georgia
  - Meridian Clinical Research-(Savannah Georgia) - Platinum - PPDS, Savannah, Georgia
  - Clinical Research Atlanta - Headlands - PPDS, Stockbridge, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Olivo Medical and Wellness Center, Chicago, Illinois
  - DM Clinical Research, River Forest, Illinois
  - Velocity Clinical Research, Valparaiso, Indiana
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC - El Dorado - PPDS, El Dorado, Kansas
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Alliance for Multispecialty Research LLC, East Wichita, Wichita, Kansas
  - Michael W Simon MD, PSC, Lexington, Kentucky
  - Velocity Clinical Research - Lafayette - PPDS, Lafayette, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Great Lakes Research Institute, Southfield, Michigan
  - DM Clinical Research, Southfield, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Sundance Clinical Research - ERN - PPDS, St Louis, Missouri
  - Meridian Clinical Research (Grand Island, Nebraska), Grand Island, Nebraska
  - Meridian Clinical Research (Norfolk-Nebraska) - Platinum - PPDS, Norfolk, Nebraska
  - Quality Clinical Research - ClinEdge - PPDS, Omaha, Nebraska
  - Meridian Clinical Research-(Omaha Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - Meridian Clinical Research, LLC (Lincoln Nebraska), Omaha, Nebraska
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Meridian Clinical Research, Binghamton, New York
  - Velocity Clinical Research, East Syracuse, New York
  - Meridian Clinical Research, Endwell, New York
  - Lucas Research, Morehead City, North Carolina
  - Lucas Research, New Bern, North Carolina
  - Meridian Clinical Research, Cincinnati, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Benchmark Research - Austin - PPDS, Austin, Texas
  - Tekton Research - Texas - Platinum - PPDS, Austin, Texas
  - ACRC Trials - Hunt - PPDS, Carrollton, Texas
  - Velocity Clinical Research - Austin - PPDS, Cedar Park, Texas
  - Cedar Health Research - Fort Worth - PPDS, Dallas, Texas
  - Benchmark Research - Fort Worth - HyperCore - PPDS, Fort Worth, Texas
  - Ventavia Research Group, Houston, Texas
  - DM Clinical Research - Texas Center For Drug Development - ERN - PPDS, Houston, Texas
  - ACRC Trials - Legacy Medical Village Headquarters, Plano, Texas
  - ACRC Trials, Plano, Texas
  - Victoria Clinical Research Group, Victoria, Texas
  - Tanner Clinic, Layton, Utah
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Health Research of Hampton Roads Inc. - Newport News, Newport News, Virginia
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia
  - Clinical Research Partners LLC - Richmond - ERN - PPDS, Richmond, Virginia